CLINICAL TRIAL: NCT00850902
Title: Application of a Different Incubator Humidity Strategy at Birth to Decrease Morbidity and Mortality in Extremely Low Birth (1000 g or Less) Infants
Brief Title: Humidity Strategy to Decrease Morbidity and Mortality in Extremely Low Birth Weight Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Fahad Medical City (Other Government)
Responsible Party: Jasim Anabrees, King Fahad Medical City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-049
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2009-03-10 (Estimated); Status verified 2009-03

CONDITIONS: Extremely Low Birth Weight
Keywords: ELBW; Humidity; BPD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate Humidity (MH) (Active Comparator)
  Interventions: Other: Moderate Humidity
- High Humidity (Experimental)
  Interventions: Other: High Humidity (HH)

INTERVENTIONS:
Other: High Humidity (HH) — High Humidity Level
  Arms: High Humidity
Other: Moderate Humidity — Moderate Humidity Level
  Arms: Moderate Humidity (MH)

SUMMARY:
The purpose of this study is to apply a different incubator humidity strategy at birth to decrease morbidity and mortality in extremely low birth (1000 g or less) infants.

ELIGIBILITY:
Inclusion Criteria:

* Inborn Premature Infants with weight ≤ 1000 g at birth

Exclusion Criteria:

* Outborn infants.
* Failure to obtain parental consent for the study.
* Congenital malformations likely to affect life expectancy or neurosensory development.
* Unlikely to be available for follow up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Death prior to discharge or Bronchopulmonary Dysplasia (BPD) defined as oxygen requirement at 36 weeks postmenstrual age. | 36 weeks postmenstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Jasim Anabrees, Principal Investigator — King Fahad Medical City